CLINICAL TRIAL: NCT06816771
Title: Evaluation of Efficacy and Safety of Pazopanib Combined with TGI/CIV(nab⁃Paclitaxel+ Gemcitabine + Ifosfamide/cyclophosphamide +Irinotecan + Vinorelbine) in the Treatment for Children or Adolescents with Recurrent/refractory Rhabdomyosarcoma--an Open-label, Single-arm, Single-cente,phase II Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Pazopanib in Combination with TGI/CIV for Recurrent or Refractory Rhabdomyosarcoma in Children or Adolescents
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jingfu Wang, MD,Principal Investigator, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-413-02
Record Dates: First submitted 2025-02-03; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Rhabdomyosarcoma, Recurrent, Refractory
Keywords: rhabdomyosarcoma; pediatric
MeSH Terms: conditions — Rhabdomyosarcoma; Recurrence | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): The participant take pazopanib once daily orally in combination with a total of 2 cycles(6 weeks) of TGI chemotherapy(nab⁃Paclitaxel+ gemcitabine + ifosfamide)/CIV(cyclophosphamide +Irinotecan + vinorelbine).Each cycle of TGI/CIV chemotherapy will last for 3 weeks, TGI will be given in cycle 1 and CIV will be given cycle 2 . At week 6, the participant will have scans and tests to reevaluate the tumor's response to the treatment. The participant will receive an additional 6 weeks (2 cycles) of the same chemotherapy in the absence of disease progression or unacceptable toxicity. After 4 cycles of chemotherapy, The investigator will re-evaluate the tumor again at week 12 and the patient will undergo other treatments(chemotherapy, radiation, surgery, etc.), but will be closely watched for any signs of tumor recurrence or progression.
  Interventions: Drug: pazopanib; Drug: TGI chemotherapy; Drug: CIV chemotherapy

INTERVENTIONS:
Drug: pazopanib — Given PO The dosage will be determined according to the participant's body surface area, with body surface area less than 0.75, 1 tablet, and 2 tablets for body surface area greater than 1. 0.75-1,1.5 tablets.
Drug: TGI chemotherapy — TGI chemotherapy (nab⁃Paclitaxel+ gemcitabine + ifosfamide)
Drug: CIV chemotherapy — CIV chemotherapy (cyclophosphamide +Irinotecan + vinorelbine)

SUMMARY:
To evaluate the efficacy and safety of pazopanib combined with TGI/CIV chemotherapy in children and adolescents with recurrent or refractory rhabdomyosarcoma.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed rhabdomyosarcoma (RMS).
2. Patients diagnosed with recurrent/refractory RMS based on clinical diagnostic criteria. Recurrence is defined as disease recurrence confirmed after achieving complete remission and completing at least one line of standard treatment; refractory is defined as disease progression as per the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) after at least four cycles of first-line chemotherapy.

   First-line standard treatment can refer to the "Diagnosis and Treatment Guidelines for Rhabdomyosarcoma in Children and Adolescents (2019 Edition)".
3. Patients must have measurable lesions as per RECIST 1.1 criteria.
4. Age ≥ 2 years and ≤ 18 years, with no gender restrictions.
5. Karnofsky Performance Scale (KPS) score of 70-100% (> 12 years) or Lansky Performance Scale score of 70-100% (≤ 12 years).
6. Expected survival time ≥ 12 weeks.
7. Before initiating any project-related procedures, the parents/guardians of the child or adolescent subjects must be able to understand, consent, and sign the informed consent form (ICF) and applicable assent form; the subjects must be able to express consent with the consent of their parents/guardians (if applicable).
8. Adequate organ and bone marrow function, defined as follows:

Bone marrow function:

1. Absolute neutrophil count (ANC) ≥ 1.5×109/L (≥ 0.5×109/L if bone marrow metastasis)
2. Platelet count ≥ 100×109/L (≥ 75×109/L if bone marrow metastasis) Hb ≥ 65 g/L (blood transfusion is allowed)
3. Hematopoietic growth factors: Treatment should be initiated at least 14 days after the last administration of long-acting growth factors or 1 day after the last administration of short-acting growth factors. renal function

1) Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) 2) If serum creatinine > 1.5 ULN, creatinine clearance rate > 70 ml/min/1.73 m² Liver function

1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver metastasis)
2. Total bilirubin ≤ 1.5 times ULN Cardiac function

1) Echocardiography LVEF ≥ 50%; 2) No severe cardiac rhythm or conduction abnormalities on electrocardiogram.

Exclusion criteria:

1. Received any of the following treatments within 2 weeks before treatment: radiotherapy, chemotherapy, or molecular targeted therapy for tumors; other investigational drugs; or live attenuated vaccines.
2. Patients who have received anti-angiogenic targeted drugs such as apatinib, pazopanib, sunitinib, sorafenib, bevacizumab, imatinib, crizotinib, famitinib, anlotinib, regorafenib, endostatin, etc. within the past 3 months.
3. Central nervous system metastasis.
4. A history of thrombosis within 3 months before enrollment and anticoagulation treatment for less than 6 weeks.
5. Known bleeding tendency, significant clinical bleeding symptoms within 3 months before treatment or definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ or above, vasculitis, etc.; or thrombotic events within 6 months before treatment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.; or need long-term anticoagulation treatment with warfarin or heparin, or need long-term antiplatelet treatment (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day).
6. Uncontrolled hypertension and proteinuria in the recent period. And cannot be well controlled by antihypertensive drugs (infants > 100/60 mmHg, preschool children (< 6 years old) > 110/70 mmHg, school-age children (6-12 years old) > 120/80 mmHg, adolescents and adults > 140/90 mmHg).
7. Use of antiepileptic drugs.
8. Long-term unhealed wounds, ulcers or fractures, major surgery within 28 days before enrollment or minor surgery within 7 days, abdominal fistula, gastrointestinal perforation.
9. Uncontrolled severe infection.
10. The presence of active heart disease within 6 months before treatment, including myocardial infarction, severe/unstable angina, etc. Poorly controlled arrhythmias with left ventricular ejection fraction < 50% on echocardiography (including QTcF intervals >450 ms in men and >470 ms in women).
11. Any other malignancy was diagnosed within 3 years before treatment.
12. Known allergy to the study drug or any of its excipient.
13. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B surface antigen positive and HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA above the detection limit of the assay).
14. According to the judgment of the researchers, patients with large tumors, easy to rupture and bleeding, and bleeding caused by tumor retraction are at high risk.
15. Concomitant medical conditions (e.g., poorly controlled hypertension, severe diabetes, neurological or psychiatric conditions, etc.) or any other condition that, in the investigator's judgment, could seriously endanger the safety of the subject, confound the study results, or interfere with the completion of the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Up to 4 cycles of chemotherapy (each cycle is 21 days)
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 4 cycles of chemotherapy (each cycle is 21 days)
  Refers to the percentage of patients with confirmed complete response, partial response, and disease stability in patients with evaluable efficacy
Incidence of adverse events | Up to 4 cycles of chemotherapy (each cycle is 21 days)
  Use NCI-CTCAE version 5.0 for classification and grading

CONTACTS AND LOCATIONS:
Overall Officials: Jingfu Wang, MD, Study Chair — Shandong Cancer Hospital and Institute
Locations (1):
- No. 440 Jiyan Road, Jinan City, Shandong Province, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No